CLINICAL TRIAL: NCT03073057
Title: Pharmacokinetic Pilot Study Comparing Three Formulations of Budesonide/Formoterol Easyhaler 160/4.5 Microg/Inhalation and Symbicort Turbuhaler: A Randomised, Open, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Study to Compare Absorption of Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3103014
Record Dates: First submitted 2016-02-15; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2016-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Charcoal and Budesonide/formoterol Easyhaler A (Experimental): 160/4.5microg/inhalation Charcoal
  Interventions: Drug: Budesonide/formoterol; Other: Charcoal
- Charcoal and Budesonide/formoterol Easyhaler B (Experimental): 160/4.5microg/inhalation Charcoal
  Interventions: Drug: Budesonide/formoterol; Other: Charcoal
- Charcoal and Budesonide/formoterol Easyhaler C (Experimental): 160/4.5microg/inhalation Charcoal
  Interventions: Drug: Budesonide/formoterol; Other: Charcoal
- Charcoal and Symbicort Turbuhaler (Active Comparator): 160/4.5microg/inhalation Charcoal
  Interventions: Other: Charcoal; Drug: Symbicort Turbuhaler

INTERVENTIONS:
Drug: Budesonide/formoterol — 2 inhalations as a single dose
  Other Names: Budesonide/formoterol 160/4.5microg
  Arms: Charcoal and Budesonide/formoterol Easyhaler A; Charcoal and Budesonide/formoterol Easyhaler B; Charcoal and Budesonide/formoterol Easyhaler C
Other: Charcoal
Drug: Symbicort Turbuhaler — 2 inhalations as a single dose
  Other Names: Symbicort Turbuhaler 160/4.5 microg
  Arms: Charcoal and Symbicort Turbuhaler

SUMMARY:
The purpose of this study is to compare Budesonide/formoterol Easyhaler test products with the marketed product Symbicort Turbuhaler in terms of the drug absorbed into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Body mass index > 19 and < 30kg/m2, weight at least 50 kg
* Good general health ascertained by detailed medical history, and laboratory and physical examinations

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during a study.
* Known hypersensitivity to the active substance(s) or the excipient of the drug
* Pregnant and lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cmax of plasma budesonide and formoterol | within 24 hours
AUCt of plasma budesonide and formoterol | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Iissa Kivisto, Study Director — Orion Corporation, Orion Pharma; Leena Mattila, MD, Principal Investigator — Orion Pharma, Clinical Pharmacology Unit, Espoo, Finland
Locations (1):
- Orion Pharma, Clinical Pharmacology Unit, Espoo, Finland